CLINICAL TRIAL: NCT07150910
Title: Comparison of the Clinical Efficacy and Patient Acceptance of Interdental Brushes and Rubber Bristles Interdental Cleaners in Patients With Gingivitis: A Randomized Controlled Trial
Brief Title: Clinical Efficacy and Patient Acceptance of Interdental Brushes and Rubber Bristles in Patients With Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Umut BALLI, Associate professor, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/15
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2021-09

CONDITIONS: Oral Hygiene

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IDB (Active Comparator): The interdental brush(IDB) used in the study (TePe® Interdental Brushes Original) is available in nine different sizes, color-coded according to brush diameter, ranging from 0.4 mm to 1.5 mm
  Interventions: Behavioral: Interdental brush
- RBIC (Active Comparator): The rubber bristles interdental cleaner features soft, flexible, and tapered synthetic rubber bristles.
  Interventions: Behavioral: Rubber bristles interdental cleaner

INTERVENTIONS:
Behavioral: Interdental brush — In accordance with the manufacturer's recommendations, the IDBs were stated to be suitable for multiple uses. Participants were advised to replace the IDB once the bristles lost their shape or if the metal wire became damaged.
  Arms: IDB
Behavioral: Rubber bristles interdental cleaner — Two sizes were selected for the study: XS/S - Orange, designed for narrow and very narrow interdental spaces, and M/L - Turquoise, suitable for medium to large spaces. Since the tested RBICs were designed by the manufacturer for single use, participants were instructed to use a new RBIC at each application.
  Arms: RBIC

SUMMARY:
The primary aim of this clinical study is to compare the effects of IDBs and RBICs on the removal of microbial dental plaque and gingival bleeding in patients with gingivitis. Secondarily, the study aims to assess participants' satisfaction and attitudes toward using these tools.

DETAILED DESCRIPTION:
This study involved 40 systemically healthy, right-handed, non-smoking patients aged 18-35 with gingivitis and no prior experience with interdental cleaning tools. Inclusion criteria required a probing depth ≤3mm, a full-mouth bleeding on probing score ≥20%, at least 20 natural teeth, and a minimum of four evaluable interproximal sites per quadrant compatible with both test devices. Key exclusion criteria were severe gingivitis, attachment loss, systemic diseases, recent antibiotic use, and pregnancy.

Participants received standardized toothpaste, a toothbrush, and training in the modified Stillman brushing technique. Following a 2-week training phase on product use and a professional prophylaxis, they refrained from interdental cleaning for 3 days to allow plaque accumulation for baseline assessments (T-QHPI for plaque, PBI for gingival bleeding).

The study employed a split-mouth design. After baseline, one side of the mouth was assigned an interdental brush (IDB - TePe® Original, sizes 0.4-1.5mm) for daily use, and the contralateral side was assigned a rubber bristle interdental cleaner (RBIC - TePe EasyPick™, XS/S or M/L size). Participants were instructed on proper insertion and technique for each device.

After two weeks of use, clinical indices were re-recorded by a blinded examiner. Additionally, participants completed a questionnaire assessing their satisfaction with various aspects of the products (cleaning capacity, accessibility, ease of use, overall satisfaction, willingness to reuse, and pain experienced during use).

ELIGIBILITY:
Inclusion Criteria:

* probing sulcus depth ≤ 3 mm and full-mouth bleeding on probing (BOP) score ≥ 20%
* presence of at least 20 natural teeth (excluding third molars), with a minimum of five teeth per quadrant
* at least four evaluable interproximal sites without crowns or restorations in each quadrant of the maxilla and mandible
* compatibility of both interdental cleaning devices with a minimum of four interproximal spaces per quadrant
* no prior experience with interdental cleaning tools
* willing to participate
* capable of understanding and complying with the study procedures and instructions.

Exclusion Criteria:

* smoking
* presence of severe gingivitis or clinical attachment loss
* systemic diseases
* use of antibiotics within the past three months
* use of anticoagulant medications or mouthwashes
* pregnancy or lactation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Plaque Levels | 2 weeks
  Plaque levels were assessed using the Turesky modification of the Quigley and Hein Plaque Index (T-QHPI). In each participant, dental plaque was disclosed using Mira-2-Ton® (Duisburg, Germany) and then rinsed with water (10 mL for 10 seconds). The stained plaque was scored on a scale from 0 to 5 as follows: 0 = no plaque; 1 = separate flecks of plaque at the cervical margin; 2 = a thin continuous band of plaque (up to 1 mm) at the cervical margin; 3 = plaque covering not more than one-third of the tooth surface; 4 = plaque covering more than one-third but not more than two-thirds of the tooth surface; 5 = plaque covering more than two-thirds of the tooth surface.
Gingival condition | 2 weeks
  Gingival condition was evaluated using the Papillary Bleeding Index (PBI) introduced by Saxer and Mühlemann. Measurements were performed by a blinded, calibrated examiner on four sites per tooth (mesiobuccal, distobuccal, mesiolingual, and distolingual). A manual UNC-15 mm periodontal probe (Hu-Friedy, Chicago, IL, USA) was carefully inserted into the gingival sulcus at the base of the papilla on the mesial side and moved coronally toward the tip of the papilla. The same procedure was repeated on the distal aspect. Bleeding severity was scored on a scale from 0 to 4: 0 = no bleeding; 1 = a single discreet bleeding point visible after 20 seconds; 2 = a fine line of blood or multiple bleeding points in the papilla; 3 = blood filling the entire interdental space; 4 = profuse bleeding that overflows from the interdental area

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No